CLINICAL TRIAL: NCT06992687
Title: A Phase I/II, Open-Label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of HB0052 in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety and Efficacy of HB0052 in Patients With Advanced Solid Tumors
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other); Zhejiang Cancer Hospital (Other); Shandong Cancer Hospital and Institute (Other); Hunan Cancer Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB0052-01
Record Dates: First submitted 2025-04-23; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumors
Keywords: HB0052

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HB0052 (Experimental): IV every 3 weeks (q3w)
  Interventions: Drug: HB0052 Injection

INTERVENTIONS:
Drug: HB0052 Injection — An antibody- drug conjugate (ADC) that targets CD73 with SN38 as the payload

SUMMARY:
To evaluate the safety and tolerability of HB0052 in patients with advanced solid tumors

DETAILED DESCRIPTION:
To determine the maximum tolerated dose (MTD) or dose-limiting toxicity（DLT）or optimal biological dose (OBD) and/or the recommended Phase 2 doses (RP2Ds) for HB0052.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years
* The subject is able to understand and willing to sign the ICF and is willing and able to comply with all study procedures.
* Patients with known UGT1A1 genotype determination results or is willing to accept UGT1A1 genotype determination test.
* For subjects in phase 2 studies, previous tumor biopsy specimens or fresh tumor biopsy specimens is required.
* Phase I: Patients with histologically or cytologically confirmed locally advanced, recurrent, or metastatic solid tumors (or clinically diagnosed hepatocellular carcinoma) that failed (progressed on or are intolerant of) all standard therapies known to provide clinical benefit [These solid tumors include but not limited to: pancreatic, colorectal, ovarian, breast, lung, head and neck, prostate, renal cancer and sarcoma, etc.].
* Phase II: Patients who have had at least one prior systemic therapy and has progressed, and might benefit from the study drug in the Investigator's judgment, and have the following histological types (The types of tumors and the number of treatment lines may be adjusted based on phase I results and /or SRC discussions):

  a.Pancreatic cancer cohort: i.Histologically or cytologically confirmed unresectable, locally advanced or metastatic pancreatic ductal adenocarcinoma; b.Endometrial carcinoma cohort: i.advanced/unresectable, recurrent, or metastatic endometrial carcinoma, or recurrent, metastatic histologically uterine serous papillary carcinoma (USPC) with measurable disease.

  c.Gastric and GEJ adenocarcinoma cohort: i.Histologically or cytologically confirmed locally advanced unresectable or metastatic gastric and GEJ adenocarcinoma ii.HER2 low expression and negative for claudin 18.2 d.RCC cohort: i.Pathologically (histologically or cytologically) proven of locally advanced unresectable or metastatic renal cell carcinoma.

  e.HCC cohort: i.inoperable locally advanced, recurrent, or metastatic HCC ii.Patients with Child-Pugh grade A liver function

  f.Other histologically confirmed unresectable, locally advanced or metastatic advanced solid tumor cohort(s): Tumor specific type that demonstrated partial response to HB0052 in the dose escalation phase.
* At least one measurable lesion as per RECIST v. 1.1 defined as non-nodal lesions having at least one dimension with a minimum size of 10 mm in the longest diameter by CT or MRI scan or ≥15 mm in short axis for nodal lesions. Radiographic disease assessment at baseline can be performed up to 28 days prior to the first dose.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
* Life expectancy ≥12 weeks.
* Patients with active hepatitis B virus (HBV) without active disease (HBV DNA titer <1000 cps/mL or 200 IU/mL), or who are cured of hepatitis C virus (HCV) with a negative HCV RNA test may be enrolled at the investigator's discretion.
* Patients with known human immunodeficiency virus (HIV) infection and a cluster of differentiation 4 (CD4) count that is tested or documented to be ≥350 cells/mm3 within 12 months before study screening.
* Adequate organ function as defined by the following criteria:
* Women of childbearing potential must confirm a negative serum pregnancy test within 3 days prior to the initiation of study treatment and begin use of an effective birth control directly after testing negative for pregnancy; Fertile patients and their partners must agree to use acceptable contraception for the duration of study drug use and for 120 days after the last administration of study treatment.
* Recovery to Grade 0-1 from adverse events (AEs) related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, and endocrinopathies controlled with hormone replacement therapy.

Exclusion Criteria:

* Concurrent malignancy < 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma. Patients with prostate cancer that is under active surveillance are eligible.
* Patients with Gilbert's disease
* Patients with a history of COPD or other severe respiratory disease in the 6 months before screening
* Patients with active ≥ grade 2 anorexia, nausea or vomiting.
* Patients with a history of intestinal obstruction or perforation in the 6 months before screening
* Patients with grade 3 or higher toxicity due to irinotecan use
* Patients with reduced UGT1A1 activity or who are predisposed to or have a history of chronic diarrhea.
* Have clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain or meningeal metastases may participate and be eligible for treatment provided they are stable and asymptomatic. Patients with asymptomatic brain or meningeal metastasis or patients who are symptomatically stable after treatment and are on ≤ 10 mg/d prednisone or equivalent are eligible.
* Cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction (MI), unstable angina, or New York Heart Association (NYHA) class III or IV heart failure occurred within 6 months before study admission；Has an average of Fredericia's formula-QT corrected interval (QTcF) prolongation to > 450 millisecond (ms) in males and > 470 ms in female; malignant arrhythmia < 3 months of study entry (judged by the Investigator). Has a history of cardiomyopathy or myocarditis. Patients with rate-controlled arrhythmias may be eligible for study entry at discretion of the Investigator.
* Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening. The following exceptions can be included: hypothyroidism, vitiligo, Graves' disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
* Patients who have previously received allogeneic stem cell or solid organ transplantation.
* History of severe allergic reactions, Grade 3-4 allergic reactions to treatment with another monoclonal antibody or known to be allergic to protein drugs or recombinant proteins or excipients in HB0052 drug formulation.
* History of Gr3-4 immune-related adverse events (irAEs) or irAEs requiring discontinuation of prior therapies, (except for Gr3 endocrinopathy that is managed with hormone replacement therapy).
* Continuous systemic corticosteroids administration in a dose equivalent to 10 mg/day or more of prednisone or prednisone-equivalent or other immunosuppressants for 5 days or more within 2 weeks before screening. The following exceptions are allowed: the use of corticosteroids in a short course (within one week) to administration topical, intraocular, intraarticular, intranasal, or inhaled are allowed.
* Have received or will receive a live vaccine within 4 weeks prior to the first dose.
* Any of the following infections

  1. Positive COVID-19 qRT-PCR or rapid screening test during screening; can be eligible one week after COVID-19 test becomes negative.
  2. Patients with active tuberculosis (TB) who are receiving anti-TB treatment or who received anti-TB treatment within 1 year prior to screening.
  3. Active bacterial infection unresolved less than 2 weeks prior to first dose of study drug
* Prior treatment with agents targeting CD73 or A2AR.
* Anticancer therapy < 5 half-lives or 4 weeks (whichever is shorter) prior to study entry;; CYP3A4 inhibitors and/or inducers therapy or OATP inhibitors therapy < 3 half-lives or 4 weeks (whichever is shorter) prior to study entry; palliative radiotherapy to a single area < 2 weeks prior to study screening is permitted. Measurable lesions cannot be previously irradiated unless they have demonstrated growth after radiation therapy (RT).
* Major surgery or chemotherapy/ interventional therapy/radiation therapy/ablation therapy < 4 weeks prior to the first dose and those who have experienced significant trauma or require elective major surgery during the study period (needle biopsy, needle drainage, bronchoscopy or venous cannulation allowed enrolling.)
* Patients who have participated in any clinical trial of a drug, biologic or medical device within 4 weeks prior to the first dose.
* Psychiatric, psychological, familial condition or geographical location that, in the judgment of the Investigator, may interfere with the planned staging, treatment and follow-up and affect patient's compliance or place the patient at high risk from treatment.
* Other conditions which would make it inappropriate for the patient to participate as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 12 Months
  Number of participants with a Dose Limiting Toxicity (DLT) [ Time Frame: During the first 21 days ]DLTs will be assessed during the first 21 days of treatment for dose-escalation phase and are defined as toxicities that meet pre defined severity criteria, and assessed as having a suspected or definite relationship to study drug
MTD | Up to 24 Months
  MTD or OBD and/or RP2D.

SECONDARY OUTCOMES:
AUC | Up to 24 Months
  Area Under concentration-time Curve (AUC)
Cmax | Up to 24 Months
  Maximum serum concentration (Cmax)
Tmax | Up to 24 Months
  Half-life time of maximum concentration

OTHER OUTCOMES:
ORR assessment in dose-escalation phase | Up to 24 Months
  Overall response rate (ORR) as measured by RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No